CLINICAL TRIAL: NCT06426992
Title: Evaluation of Clinical Effectiveness of Microwave Ablation Using Starwave Microwave Generator for Small Liver Malignancies: A Prospective Single Center Study
Brief Title: Clinical Effectiveness of Microwave Ablation Using Starwave Microwave Generator for Hepatic Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2402-111-151
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Liver Malignant Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with malignant liver tumors (Experimental): Following the existing procedure of our institute, we aim to treat the tumor by applying up to 150W of microwaves within the tumor using a StarWave microwave generator and a 13-gauge antenna under fusion ultrasound guidance. If necessary, the antenna is reinserted 1-2 times to create sufficient ablation lesions until an echogenic band of 5-10mm is formed around the tumor and its periphery, implementing overlapping microwave ablation (MWA). Afterward, the antenna is removed while applying microwave energy to prevent bleeding.
  Interventions: Procedure: Microwave ablation

INTERVENTIONS:
Procedure: Microwave ablation — Following the existing procedure of our institute, we aim to treat the tumor by applying up to 150W of microwaves within the tumor using a StarWave microwave generator and a 13-gauge antenna under fusion ultrasound guidance. If necessary, the antenna is reinserted 1-2 times to create sufficient ablation lesions until an echogenic band of 5-10mm is formed around the tumor and its periphery, implementing overlapping microwave ablation (MWA). Afterward, the antenna is removed while applying microwave energy to prevent bleeding.

SUMMARY:
The purpose of this study is to determine the technical success rate of creating a safety margin of 5 mm or more including the tumor by performing image-guided percutaneous microwave thermal therapy using a microwave generator and antenna developed by StarMed for the treatment of small liver cancer and the 1-year local recurrence rate based on follow-up imaging tests.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class A or B
* Patients with suspected hepatocellular carcinoma or residual/recurrent hepatocellular carcinoma of 4 cm or less on MDCT, CEUS, or MRI performed within the last 60 days or Patients with suspected metastatic liver cancer of 4 cm or less on MDCT, CEUS, or MRI performed within the last 60 days, for whom microwave thermal ablation is being considered

Exclusion Criteria:

* In cases where there are three or more malignant liver tumors
* When the maximum size of the tumor exceeds 4 cm
* Diffuse infiltrative type of cancer with unclear tumor boundaries
* When the tumor is adhered to the central hepatic portal vein, hepatic vein, or bile duct by 5 mm or more
* Severe liver failure (Child-Pugh Class C)
* In cases of vascular invasion by malignant liver tumors
* Severe coagulopathy (platelet count below 50,000/mm³ or INR prolonged by more than 50%)
* In cases of multiple extrahepatic metastases
* Situations where it is highly unlikely to obtain appropriate data for research purposes

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | Immediately after ablation
  Technical success addresses whether the index tumor was treated according to a predefined protocol and entirely covered by the ablation zone.
Local tumor progression rate | 12 months after ablation
  Local tumor progression, defined as the appearance of tumor foci at the margin of the ablation zone after the attainment of treatment success

SECONDARY OUTCOMES:
Complication after ablation | Immediately, 1 month, 3 months, 6 months, 9 months, and 12 months after radiofrequency ablation
  Post ablation complications were defined as problems noted within 1 month after MWA as well as additional complications identified on follow-up imaging and judged to be likely caused by ablation.
Recurrence-free survival | 12 months after ablation
  Recurrence-free survival was defined as the interval between ablation and the date of any type of recurrence or the last follow-up date if there was no recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea